CLINICAL TRIAL: NCT04796675
Title: Safety and Efficacy of Cord Blood Derived Anti-CD19 CAR-Engineered NK Cells for Relapsed/Refractory B Lymphoid Malignancies: a Single-center, Open-label, Single-arm Clinical Study
Brief Title: Cord Blood Derived Anti-CD19 CAR-Engineered NK Cells for B Lymphoid Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Shanghai Simnova Biotechnology Co.,Ltd. (Industry)
Responsible Party: Principal Investigator, MEI HENG, Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-NK-CD19 cells
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Non Hodgkin's Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Cyclophosphamide + CAR-NK-CD19 Cells (Experimental): Patients will received lymphodepletion with fludarabine (30 mg/kg) and cyclophosphamide (300 mg/kg) on day -5, -4, and -3, followed by one infusion of CAR-NK-CD19 cells on day 0. The study will be divided into three groups: Acute Lymphocytic Leukemia, Chronic Lymphocytic Leukemia, and Non Hodgkin's Lymphoma. Doses of 0.01×10^7, 0.1×10^7, 1.0×10^7 CAR+ T cells (with an allowance of ±20%) will be tested in each group in the 3+3 dose-escalation study. Each dose group has 3 patients. If no dose-limited toxicity (DLT) emerges in the group, then the subsequent higher dose will be used in the next group. If DLT emerges in a single subject in any dose level, 3 more subjects will be enrolled to the same dose level. The maximum dose could be extended.
  Interventions: Drug: Fludarabine + Cyclophosphamide + CAR-NK-CD19 Cells

INTERVENTIONS:
Drug: Fludarabine + Cyclophosphamide + CAR-NK-CD19 Cells — fludarabine 30 mg/kg on day -5, -4, and -3; cyclophosphamide 300 mg/kg on day -5, -4, and -3; CAR-NK-CD19 Cells on day 0.

SUMMARY:
This is a single-center, open-label, single-arm study to evaluate the primary safety and efficacy of anti-CD19 chimeric antigen receptor(CAR)-modified NK cells(CAR-NK-CD19) in patients with relapsed or refractory hematological malignancies.

DETAILED DESCRIPTION:
Anti-CD19 chimeric antigen receptor (CAR) T-cell therapy has shown remarkable clinical efficacy in B-cell cancers. However, CAR T cells can induce substantial toxic effects, and the manufacture of the cells is complex. Natural killer (NK) cells that have been modified to express an anti-CD19 CAR have the potential to overcome these limitations.

Cord blood(CB) derived NK cells from healthy donor are the source for production of CAR-NK-CD19 cells. CB derived NK cells are purified and transduced with a retroviral vector encoding the anti-CD19 CAR and interleukin-15.

This is an investigational study. The objectives are to evaluate the safety and efficacy of CAR-NK-CD19 cells in patients with CD19+ B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years;
2. Eastern Cooperative Oncology Group score≤ 3;
3. Diagnosed as CD19+ B-cell hematological malignancies, including acute lymphoblastic leukemia, chronic lymphocytic leukemia and Non Hodgkin's lymphoma.
4. Patients must relapse or be refractory after at least two lines of therapy.
5. Patient's main organs functioning well:

   A. Liver function: alanine aminotransferase/aspartate aminotransferase < 2.5 times the upper limit of normal (ULN) and total bilirubin≤ 1.5 times ULN; B. Renal function: Creatinine clearance rate ≥ 60ml/min. C. Pulmonary function: Indoor oxygen saturation ≥ 95%. D. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥50%, no clinically-significant ECG findings.
6. Negativity of blood pregnancy test for woman, and participants use effective methods of contraception until last follow-up.
7. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.

Exclusion Criteria:

1. Investigators judge the patients with gastrointestinal lymph node and/or central nervous system involvement who may be at high-risk of receiving CAR-NK-CD19 cell treatment.
2. Patients with graft-versus-host reaction and need immunosuppressive agents, or patients with autoimmune diseases.
3. Systemic steroids are used within 5 days before apheresis.
4. Drugs to stimulate the production of bone marrow hematopoietic cells are used within 5 days before apheresis.
5. Patients receive cytotoxic chemotherapy or radiotherapy within 21 days before enrollment(Tyrosine kinase inhibitors or other targeted therapies can be used two weeks before lymphodepleting chemotherapy).
6. History of epilepsy or other central nervous system diseases.
7. Participants with other active malignancies (except non-melanoma skin cancer and cervical cancer) within five years.
8. Known HIV positive patients.
9. Patients with active infections, including active replication of hepatitis B or active hepatitis C.
10. Patients receive any antitumor treatments within 4 weeks before enrollment, and the toxicity related to previous treatments don't return to < 1 level at enrollment (except for low grade toxicity such as alopecia).
11. Major surgery in the past 4 weeks.
12. Non-compliant patients.
13. Anticoagulants are being used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-04-10 (Estimated); Primary Completion 2023-03-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | within 2 years after infusion
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Overall response rate(ORR) of administering CAR-NK-CD19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | within 2 years after infusion
  ORR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Complete response rate(CRR) of administering CAR-NK-CD19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | within 2 years after infusion
  CRR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Progress-free survival(PFS) of administering CAR-NK-CD19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | within 2 years after infusion
  PFS will be assessed from CAR T cell infusion to death or last follow-up (censored).
Duration of Response(DOR) of administering CAR-NK-CD19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | within 2 years after infusion
  DOR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Overall survival(OS) of administering CAR-NK-CD19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | within 2 years after infusion
  OS will be assessed from CAR T cell infusion to death or last follow-up (censored).

OTHER OUTCOMES:
In vivo expansion and survival of CAR-NK-CD19 cells | within 2 years after infusion
  Quantity of CAR-NK-CD19 CAR copies in bone marrow and peripheral blood will be determined by using quantitative polymerase chain reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hu, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu E, Marin D, Banerjee P, Macapinlac HA, Thompson P, Basar R, Nassif Kerbauy L, Overman B, Thall P, Kaplan M, Nandivada V, Kaur I, Nunez Cortes A, Cao K, Daher M, Hosing C, Cohen EN, Kebriaei P, Mehta R, Neelapu S, Nieto Y, Wang M, Wierda W, Keating M, Champlin R, Shpall EJ, Rezvani K. Use of CAR-Transduced Natural Killer Cells in CD19-Positive Lymphoid Tumors. N Engl J Med. 2020 Feb 6;382(6):545-553. doi: 10.1056/NEJMoa1910607. PMID 32023374